CLINICAL TRIAL: NCT01372241
Title: An Appalachian Cervical Cancer Prevention Project
Brief Title: Faith Moves Mountains: An Appalachian Cervical Cancer Prevention Project
Acronym: FMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nancy Schoenberg (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Nancy Schoenberg, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R01CA108696 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-13 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2011-06

CONDITIONS: Cervical Cancer
Keywords: Papanicolaou test; Cervical cancer screening; Randomized controlled trial; Faith-placed; Appalachia
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Intervention (Experimental): This group served as the treatment group for analysis of the primary outcome.
  Interventions: Behavioral: Lay health advisor visits and newsletter
- Delayed Intervention (No Intervention): This group served as a wait-list control group, eventually receiving the intervention after the treatment group completed the intervention and the primary outcomes were assessed for both groups.

INTERVENTIONS:
Behavioral: Lay health advisor visits and newsletter — The focus of the intervention was on reducing participants' self-identified barriers to obtaining Pap tests.
  Arms: Early Intervention

SUMMARY:
The purpose of this study is to determine whether a faith-placed lay health advisor intervention is effective in increasing use of Pap smears among middle-aged and older Appalachian women.

DETAILED DESCRIPTION:
Project development relied on principles of community based participatory research. Participants were recruited from faith institutions in four distressed Appalachian Kentucky counties. Investigators at the University of Kentucky worked closely with local staff who implemented study procedures in the field.

ELIGIBILITY:
Inclusion Criteria:

* Outside of cervical cancer screening guidelines at the time of study initiation
* Able to provide informed consent

Exclusion Criteria:

* History of cervical cancer
* History of hysterectomy

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 345 (Actual)
Dates: Start 2005-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants self-reporting receipt of Pap test | One month post-intervention
  This measure is obtained at multiple timepoints during the study, but as the primary outcome it will be analyzed at the timepoint one month following the Early Intervention group's completion of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Schoenberg, Ph.D., Principal Investigator — University of Kentucky; Mark Dignan, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- Faith Moves Mountains, Whitesburg, Kentucky, United States

REFERENCES:
- [Background] Schoenberg NE, Hatcher J, Dignan MB, Shelton B, Wright S, Dollarhide KF. Faith Moves Mountains: an Appalachian cervical cancer prevention program. Am J Health Behav. 2009 Nov-Dec;33(6):627-38. doi: 10.5993/ajhb.33.6.1. PMID 19320612
- [Derived] Studts CR, Tarasenko YN, Schoenberg NE, Shelton BJ, Hatcher-Keller J, Dignan MB. A community-based randomized trial of a faith-placed intervention to reduce cervical cancer burden in Appalachia. Prev Med. 2012 Jun;54(6):408-14. doi: 10.1016/j.ypmed.2012.03.019. Epub 2012 Apr 3. PMID 22498022